CLINICAL TRIAL: NCT03421210
Title: Effects of Smoking Environments on Brain Reactivity
Acronym: CameraCue3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00089183; 1R01DA038442 (NIH)
Record Dates: First submitted 2018-01-22; First posted 2018-02-05 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotine Replacement Therapy (Other): Participants will receive nicotine replacement therapy for 10 weeks after quitting smoking.
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Nicotine patch — Participants will wear nicotine patches for 10 weeks after their quit date. 21mg/d patches for 6 weeks, then step down to 14mg/d patches for 2 weeks and finally step down 7mg/d for the last 2 weeks of treatment.

SUMMARY:
The goal of this study is to evaluate correlations between brain reactivity (as assessed via functional magnetic resonance imaging (fMRI) following 24-h abstinence) and the amount of smoking in a specific location. The investigators will use ecological momentary assessment (EMA) to ask smokers to rate their exposure to, and smoking in, specific personal smoking environment cues (PSEs) over the course of 2 weeks before quitting smoking and 2 weeks after quitting smoking. The investigators propose to identify 48 regular cigarette smokers who will complete 8 visits (1 screening visit, 1 training visit, 1 camera turn-in visit, 1 fMRI session and 4 post-quit medication check sessions). Multiple methods will be used to test hypotheses about brain functioning during cue-reactivity (CR). The investigators will examine correlation between brain responses to smoking environments (minus non-smoking environments) and smoking cessation outcomes (i.e. days to lapse, days to relapse). Our EMA+Global Positioning System (GPS) analysis will primarily focus on locations where smokers smoke before and after quitting smoking. The investigators will evaluate whether EMA-assessed smoking intensity values are correlated with brain responses to these personal smoking environments.

ELIGIBILITY:
Inclusion Criteria:

1. generally healthy [(i.e. ambulatory, not currently sick)]
2. between the ages of 18 and 65
3. smoking of at least 5 cig/day of a brand delivering ≥ 0.5 mg nicotine (FTC method) for > 1 year
4. an expired carbon monoxide (CO) concentration of at least 10 ppm (to confirm inhalation) or urinary cotinine >1000 ng/mL (NicAlert = 6).
5. interest in quitting smoking within the timeframe of the experiment.
6. ability to identify 4 personal smoking and 4 personal non-smoking places.
7. right handed as measured by a three-item scale used in our laboratory
8. own a smartphone

Exclusion Criteria:

1. immediate or no desire to quit smoking;
2. inability to attend all required experimental sessions;
3. use of other tobacco products or e-cigarettes more than 9 days in the past 30 days;
4. current alcohol or drug abuse;
5. positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, and Phencyclidine(PCP)

   1. marijuana will be tested for but will not be exclusionary;
   2. participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded;
   3. participants failing the toxicology screen will be allowed to re-screen once;
6. current use of nicotine replacement therapy or other smoking cessation treatment;
7. screening systolic BP greater than 140 (participants failing for blood pressure will be allowed to rescreen once)
8. screening diastolic BP greater than 90 (participants failing for blood pressure will be allowed to rescreen once)
9. screening heart rate greater than 100 (participants failing for heart rate will be allowed to rescreen once)
10. presence of conditions contraindicated for nicotine replacement therapy (e.g., skin allergies)
11. report of significant health problems including but not restricted to (e.g. chronic hypertension, emphysema, seizure disorder, history of significant heart problems, heart disease, heart attack in the past 90 days, irregular heartbeat)
12. medical condition that may contraindicate participation in the opinion of the investigator and study physician.
13. current major psychiatric disease such as schizophrenia or schizoaffective disorder
14. currently pregnant, breast feeding or likely to become pregnant;
15. a quit attempt resulting in greater than 3 days of abstinence in the past 30 days
16. presence of conditions that would make MRI unsafe (e.g., pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine Replacement Therapy
Started | 88
Received Functional Magnetic Resonance Imaging (fMRI) | 42
Completed | 35
Not Completed | 53

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study. Those with excessive head motion or artifacts identified during QA checks were not included in analyses.
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 13
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Signal Change in Functional Magnetic Resonance Imaging (fMRI) Contrast of Parameter Estimate (COPE) Between Personal Environment Pictures Relative to Non-Personal Environment Pictures
Description: Using fMRI the investigators examined brain function during cue-reactivity. During the scan, participants viewed pictures of personal and non-personal environments.
  Contrast of parameter estimate (COPE) values for the difference between personal smoking environment pictures and non-personal smoking environment pictures were extracted from anatomically defined brain regions using FSL's featquery for analysis.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: contrast of parameter estimate (COPE)
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 32
contrast of parameter estimate (COPE) | 0.0598 (0.09454)
Statistical Analysis 1: Comparison: Nicotine Replacement Therapy; Differences in brain activation in response to personal smoking versus standard smoking cues were examined; Test type: Other; p = 0.001, t-test, 1 sided

2. Secondary Outcome: Post-Quit Craving as Measured by (Ecological Momentary Assessment) EMA Questionnaire
Description: EMA will be used to evaluate craving daily for 2 weeks after quitting. Subjects will rate their craving on a single item (How strong is your current urge to smoke?) using a scale from 1 "very slightly or not at all" to 5 "extremely".
Time Frame: 2 weeks after quitting smoking
Population: All participants with post-quit EMA data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 36
score on a scale | 2.49 (1.03)

3. Secondary Outcome: Number of Participants Experiencing Relapse
Description: Relapse defined as 7 consecutive days smoking at least 1 cigarette per day. Individuals lost to contact are presumed to have relapsed following their last visit.
Time Frame: Weeks 1, 3, 6, and 10 weeks after quitting.
Population: 42 subjects entered the quit phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 42
Participants
  Week 1 | 16
  Week 3 | 9
  Week 6 | 3
  Week 10 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks after quitting smoking
Description: Adverse events were typically identified during the administration of the Side Effects form and deemed to require followup. Other events were identified from physiological measures or by spontaneous reports during assessments.Participant's fMRI session was followed by a quit day and 10 weeks of patch use (this period included 4 follow up visits). 42 participants were scanned, 32 had usable fMRI data, 35 participants completed the entire study (all 10 weeks post quit date)
Arm/Group | Nicotine Replacement Therapy
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 21/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Replacement Therapy (N=42)
Vivid Dreams (Psychiatric disorders) | 5
Rash at Patch site (Skin and subcutaneous tissue disorders) | 4
Itching/burning at patch site (Skin and subcutaneous tissue disorders) | 8
Coughing (Respiratory, thoracic and mediastinal disorders) | 5
Irritability (Psychiatric disorders) | 8
Heart Burn (Gastrointestinal disorders) | 2
Nightmares (Psychiatric disorders) | 2
Elevated CESD score (Psychiatric disorders) | 7
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Hiccups (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion/ sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Elevated Blood Pressure (Vascular disorders) | 1
Dizzyness upon standing (Vascular disorders) | 2
Feeling Faint (Vascular disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Mouth/Throat Irritation (General disorders) | 1
Hand Numbness (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03421210/Prot_SAP_000.pdf